CLINICAL TRIAL: NCT00144040
Title: Improving Antibiotic Use in Acute Care Setting
Brief Title: Improving Antibiotic Use in Acute Care Treatment
Acronym: IMPAACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: AVA 03-239; R01 HF13915
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Respiratory Infections
Keywords: Antibiotics; Respiratory Infections; Quality Assurance, Healthcare; Professional Education; Emergency Services, Medical; Education, Patient
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Physician & patient education on appropriate antibiotic use; Procedure: Rapid C-reactive protein testing to guide antibiotic treatment

INTERVENTIONS:
Behavioral: Physician & patient education on appropriate antibiotic use
Procedure: Rapid C-reactive protein testing to guide antibiotic treatment

SUMMARY:
Purpose The emergence and rapid rise in antibiotic resistance among common bacteria are adversely affecting the clinical course and health care costs of community-acquired infections. Because antibiotic resistance rates are strongly correlated with antibiotic use patterns, multiple organizations have declared reductions in unnecessary antibiotic use to be critical components of efforts to combat antibiotic resistance. Among humans, the vast majority of unnecessary antibiotic prescriptions are used to treat acute respiratory tract infections (ARIs) that have a viral etiology. Although the rate of antibiotic prescribing for ARIs by office-based physicians in the US has decreased about 16% from its peak in 1997, the rate of antibiotic prescribing in acute care settings (eg, emergency departments and urgent care centers), which account for 1 in 5 ambulatory antibiotic prescriptions in the US, has shown only a modest decline (6%) during this period. Translation of lessons from intervention studies in office-based practices is needed to improve antibiotic use in acute care settings.

DETAILED DESCRIPTION:
Objectives:

Specific Aim 1: To evaluate the impact of a multidimensional (patient, system, clinician) intervention on appropriate antibiotic use for adults with acute respiratory tract infections-- identifying factors that influence successful translation across VA hospital and non-VA hospital acute care. Specific Aim 2: To evaluate the impact of a rapid diagnostic test for c-reactive protein on antibiotic use for adults with acute cough illness when added to a multidimensional intervention.

Methods:

We propose to conduct a randomized controlled trial of a quality improvement program consisting of physician education (educational seminar, practice guidelines, performance feedback, and decision support tools) and patient education (waiting room print and audiovisual materials) in 8 VA hospital and 8 non-VA hospital emergency departments. Non VA study sites will be identified from an existing research network of hospital emergency departments--EDNet. VA hospital sites will be selected among academically affiliated hub facilities. Phase one will involve a hospital-level randomized trial of a multidimensional intervention to translate existing evidence based guidelines for antibiotic use in ARIs vs. usual care. Simultaneously, we will validate a new CRP-based diagnostic algorithm and incorporate it into the evidence based guidelines for antibiotic use in ARIs. Phase two will involve a second hospital-level randomized trial of the new antibiotic use guidelines that incorporate the CRP-based diagnostic algorithm vs. the original guidelines. Specific endpoints include the overall success of the intervention in each phase in terms of reducing antibiotic prescribing for ARIs, improving patient outcomes and reducing resource utilization. In addition we will examin the impact of VA and non-VA organizational factors on the successful translation of various components of the intervention in both phases. Data will be collected using existing administrative data as well as on-site enrollment of subjects in prospective follow-up studies.

ELIGIBILITY:
Inclusion Criteria:

* Emergency room patient
* Selected VA or Non-VA patients
* Age 18 years or older
* Patient must have acute respiratory illness
* Patient must not have been seen in Emergency Department within 4 weeks

Exclusion Criteria:

* Patients less than 18 years of age
* Patient in Emergency Department for non-acute respiratory infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2004-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Proportion of all acute respiratory infection visits treated with antibiotics

SECONDARY OUTCOMES:
Delayed antibiotic treatment of acute respiratory infections; Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Joshua P. Metlay, MD PhD, Principal Investigator — Philadelphia VA Medical Center, Philadelphia, PA
Locations (9):
- United States (9):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

REFERENCES:
- [Result] Metlay JP, Camargo CA Jr, Bos K, Gonzales R. Assessing the suitability of intervention sites for quality improvement studies in emergency departments. Acad Emerg Med. 2005 Jul;12(7):667-70. doi: 10.1197/j.aem.2005.01.012. PMID 15995102
- [Result] Gonzales R, Camargo CA Jr, MacKenzie T, Kersey AS, Maselli J, Levin SK, McCulloch CE, Metlay JP; IMPAACT Trial Investigators. Antibiotic treatment of acute respiratory infections in acute care settings. Acad Emerg Med. 2006 Mar;13(3):288-94. doi: 10.1197/j.aem.2005.10.016. PMID 16514122
- [Result] Vanderweil SG, Pelletier AJ, Hamedani AG, Gonzales R, Metlay JP, Camargo CA Jr. Declining antibiotic prescriptions for upper respiratory infections, 1993-2004. Acad Emerg Med. 2007 Apr;14(4):366-9. doi: 10.1197/j.aem.2006.10.096. Epub 2007 Feb 12. PMID 17296803
- [Result] Aspinall SL, Metlay JP, Maselli JH, Gonzales R. Impact of hospital formularies on fluoroquinolone prescribing in emergency departments. Am J Manag Care. 2007 May;13(5):241-8. PMID 17488189
- [Result] Metlay JP, Camargo CA Jr, MacKenzie T, McCulloch C, Maselli J, Levin SK, Kersey A, Gonzales R; IMPAACT Investigators. Cluster-randomized trial to improve antibiotic use for adults with acute respiratory infections treated in emergency departments. Ann Emerg Med. 2007 Sep;50(3):221-30. doi: 10.1016/j.annemergmed.2007.03.022. Epub 2007 May 23. PMID 17509729
- [Result] Nolt BR, Gonzales R, Maselli J, Aagaard E, Camargo CA Jr, Metlay JP. Vital-sign abnormalities as predictors of pneumonia in adults with acute cough illness. Am J Emerg Med. 2007 Jul;25(6):631-6. doi: 10.1016/j.ajem.2006.11.031. PMID 17606087
- [Result] Pines JM, Hollander JE, Lee H, Everett WW, Uscher-Pines L, Metlay JP. Emergency department operational changes in response to pay-for-performance and antibiotic timing in pneumonia. Acad Emerg Med. 2007 Jun;14(6):545-8. doi: 10.1197/j.aem.2007.01.022. Epub 2007 Apr 30. PMID 17470905